CLINICAL TRIAL: NCT00118521
Title: Foot Orthotics in the Treatment of Patellofemoral Pain Syndrome: A Randomised Clinical Trial in Primary Care
Brief Title: A Clinical Study in the Use of Orthotics in Treating Pain in the Front of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2003001023NHMRC; NHMRC#301037
Record Dates: First submitted 2005-07-01; First posted 2005-07-11 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2006-09

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Anterior Knee Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Physical Therapy Modalities

INTERVENTIONS:
Procedure: Foot Orthotics
Procedure: Physiotherapy

SUMMARY:
Musculoskeletal conditions account for the third leading cause of health systems expenditure in Australia. Patellofemoral pain syndrome or pain about the knee cap is such a condition often treated in primary care. Both the individual and community are affected by this condition with an estimated 1 in 4 sufferers having problems and pain up to 20 years after first being afflicted. Importantly, it interferes with activities such as walking, jogging, gym classes and aerobics, which are often prescribed to prevent serious conditions of the heart, diabetes and obesity. Hence, it negatively impacts the health and well being of our nation.

Two popular treatment options that are commonly prescribed for the management of patellofemoral pain syndrome are physiotherapy and foot orthotics. To date, there is some evidence supporting physiotherapy, especially current best practice methods, such as a combined program of therapeutic exercise, manual therapy and kneecap taping. There is a lack of evidence for the use of orthotics in treating patellofemoral pain syndrome.

This project will conduct a randomised clinical trial to evaluate the relative benefits of orthotics as the sole treatment of patellofemoral pain syndrome and also when combined with physiotherapy. Factors associated with predicting the results of orthotic therapy will be studied to see if there are any tests that a health care practitioner can perform to provide information early on in a consultation regarding possible treatment outcomes. A cost-benefit analysis will also be conducted to calculate the relative economic merits of the treatments.

A tangible outcome of this project will be the development of clinical guidelines for the most effective method of treating patellofemoral pain syndrome in primary health care.

DETAILED DESCRIPTION:
Musculoskeletal conditions account for the third leading cause of health systems expenditure in Australia. Patellofemoral pain syndrome or pain about the knee cap is such a condition often treated in primary care. Both the individual and community are affected by this condition with an estimated 1 in 4 sufferers having problems and pain up to 20 years after first being afflicted. Importantly, it interferes with activities such as walking, jogging, gym classes and aerobics, which are often prescribed to prevent serious conditions of the heart, diabetes and obesity. Hence, it negatively impacts the health and well being of our nation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of patellofemoral pain syndrome (non traumatic origin) of at least 6 weeks duration
* Pain with at least 2 of the following activities: stair walking, jogging/running, squatting, hopping/jumping, kneeling or prolonged sitting

Exclusion Criteria:

* Concomitant injury or pathology of other knee joint structures, eg. meniscal, ligamentous etc.
* Pain in or referred from the lumbar spine and hip
* History of knee fractures, patellar dislocation/subluxation with a positive apprehension test
* Prior physiotherapy treatment (including patellar taping) within the past 12 months
* History of allergic reaction to adhesive tape
* Current or previous foot orthotic use
* Any condition of the foot that precludes orthotic therapy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176
Dates: Start 2004-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Worst and Usual Pain Visual Analogue Scale
Functional Index Questionnaire
Anterior Knee Pain Scale
Patient Perceived Treatment Effect score
Perceived Global Effect 5 Point Scale

SECONDARY OUTCOMES:
Physical activity level in previous week
Step up, step down and squat tests
Lower Extremity Functional Scale
McGill Pain Questionnaire
SF-36 Health Survey
Hospital Anxiety and Depression Scale
Patient Specific Functional Scale
Pressure pain threshold

CONTACTS AND LOCATIONS:
Overall Officials: Bill Vicenzino, PhD, Principal Investigator — The University of Queensland
Locations (1):
- Musculoskeletal Pain & Injury Research Unit, Division of Physiotherapy, The University of Queensland, Brisbane, Queensland, Australia

REFERENCES:
- [Derived] Collins NJ, Bierma-Zeinstra SM, Crossley KM, van Linschoten RL, Vicenzino B, van Middelkoop M. Prognostic factors for patellofemoral pain: a multicentre observational analysis. Br J Sports Med. 2013 Mar;47(4):227-33. doi: 10.1136/bjsports-2012-091696. Epub 2012 Dec 13. PMID 23242955
- [Derived] Collins N, Crossley K, Beller E, Darnell R, McPoil T, Vicenzino B. Foot orthoses and physiotherapy in the treatment of patellofemoral pain syndrome: randomised clinical trial. Br J Sports Med. 2009 Mar;43(3):169-71. doi: 10.1136/bmj.a1735. PMID 19270165
- [Derived] Collins N, Crossley K, Beller E, Darnell R, McPoil T, Vicenzino B. Foot orthoses and physiotherapy in the treatment of patellofemoral pain syndrome: randomised clinical trial. BMJ. 2008 Oct 24;337:a1735. doi: 10.1136/bmj.a1735. PMID 18952682
- [Derived] Vicenzino B, Collins N, Crossley K, Beller E, Darnell R, McPoil T. Foot orthoses and physiotherapy in the treatment of patellofemoral pain syndrome: a randomised clinical trial. BMC Musculoskelet Disord. 2008 Feb 27;9:27. doi: 10.1186/1471-2474-9-27. PMID 18304317